CLINICAL TRIAL: NCT01040715
Title: A Phase II, Randomized, Double-blind, Controlled Study to Evaluate the Immune Responses, Safety and Clinical Efficacy of Three Doses of Neovacs' TNF-Kinoid in Adult Patients With Rheumatoid Arthritis Who Have Relapsed Despite Anti-TNFα Biological Therapy
Brief Title: Immunogenicity and Safety of TNFa Kinoid in Rheumatoid Arthritis With Secondary Resistance to TNFa Antagonists
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNF-K-003; 2009-012041-35 (Registry Identifier: EMEA)
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; anti-drug antibodies; Rheumatoid arthritis with secondary loss of efficacy to anti-TNFa antagonists and anti-drug antibodies
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TNFa Kinoid dose 1 (Experimental)
  Interventions: Biological: TNFa Kinoid; Biological: TNF kinoid
- TNFa Kinoid dose 2 (Experimental)
  Interventions: Biological: TNFa Kinoid; Biological: TNF kinoid
- TNFa Kinoid dose 3 (Experimental)
  Interventions: Biological: TNFa Kinoid; Biological: TNF kinoid

INTERVENTIONS:
Biological: TNFa Kinoid — TNFa kinoid
Biological: TNF kinoid — IM administration 2 or 3 injections within 28 days

SUMMARY:
The objective of this trial is to demonstrate that active immunization with anti-TNFα kinoid (TNF-K) is able to induce polyclonal anti-TNFα antibodies in RA patients who were previously treated with anti-TNFα mAb but have lost susceptibility to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology (ACR) (Arnett 1988) since at least six months prior to first study product administration.
* Male or female between 18 and 70 years of age at the time of the first immunization
* Active RA disease as evidenced by a Disease Activity Score 28 (DAS 28) ≥ 3.2.
* Current or past treatment with an anti-TNF antagonist (infliximab, adalimumab,etanercept, certolizumab, golimumab).
* A wash-out period before the first administration of the study product of at least ten weeks since the last administration of certolizumab or golimumab; at least eigth weeks since the last administration of infliximab; at least four weeks since the last administration of adalimumab or etanercept
* History of positive response defined as an ACR20 or DAS 28 decrease ≥ 1.2 or by the investigator opinion with previous TNFα antagonist treatment.
* Secondary treatment failure to maximum one previous TNFα antagonist treatment as defined by:
* Investigator opinion. OR
* DAS28 increase ≥ 0.6 during the last six months. OR
* Decrease in European League Against Rheumatoid (EULAR) score.
* Written informed consent .

Exclusion Criteria:

* Treatment with non-biological DMARDs within four weeks prior to first study product administration. MTX is allowed provided it is administered at as table dosage < ou = 20 mg/week since at least 4 weeks.
* Treatment with any rheumatoid arthritis biological therapy other than TNFα antagonists at any time prior to first study product administration.
* Administration of high doses of intra-articular corticosteroids for the treatment of an acute mono-arthritis (eg knee) within 3 months prior to first study product administration. High dose of corticosteroids is defined as > 50 mg triamcinolone or equivalent.
* History of documented severe bacterial infection within 28 days prior to first immunization
* History of primary resistance or intolerance to any TNFα antagonist.
* History of or current congestive heart failure, controlled or not.
* Corticosteroids (prednisone or equivalent, < ou = 10 mg per day) are allowed if they are administered at stable dosage since at lesat 4 weeks prior to the first immunization. Inhaled and topical steroids are allowed.
* Known history of tuberculosis (TB).
* Suspicion of TB at chest X-rays at screening or within three months prior to first administration of study product.
* Suspicion of latent or active tuberculosis as defined by :
* Positive Mantoux/Purified Protein Derivative (PPD)test (> ou = 5mm induration measured 48 to 72 hours after intradermal injection of tuberculin) at screening or within 30 days prior to first administration of study product.
* and/or positive interferon-γ (IFN γ) TB diagnostic test (as measured by the ELISpot method) at screening or within three months prior to first administration of study product.
* Positive for HIV, HCV or HBV including HBsAg and anti-HBc antibodies.
* Use of any investigational or non-registered product (drug or vaccine).
* Administration of any live vaccine within three months prior to study entry
* Any confirmed or suspected immunosuppressive or immunodeficient condition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with at least a 3-fold increase in antibody response to TNFa vs baseline at day 38 | Day 38

SECONDARY OUTCOMES:
Proportion of patients with a decrease of at least 1.2 in DAS28 at month 3 vs baseline | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Durez, MD, Principal Investigator — Cliniques Universitaires St Luc
Locations (35):
- Argentina (5):
  - Centro especializado en Investigaciones Medicas (CEIM), Buenos Aires
  - Hospital Sirio Libanes, Buenos Aires
  - Hospital Italiano de Cordoba, Córdoba
  - Centro de Investigaciones Reumatologicas, San Miguel de Tucumán
  - Centro Médico Privado de Reumatología, San Miguel de Tucumán
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - Universiteit ZiekenHuis Katholiek Universiteit Leuven, Leuven
  - Universitaires Cliniques St. Luc (Mont-Godinne), Mont-Godinne
- Bulgaria (6):
  - Diagnostic and Consulting Center SV, Plovdiv
  - Military Medical Academy, Sofia
  - National Multiprofile Transport Hospital "Tzar Boris III", Sofia
  - University Hospital for Active Treatment "Sveti Ivan Rilski", Sofia
  - MBAL University Stara Zagora, Stara Zagora
  - Medical Center "Chaika" Ltd, Varna
- Chile (2):
  - "Sociedad Médica del Aparato Locomotor SA", Santiago
  - Centro de Estudios Reumatológicos- Estudios Clínicos Limitada", Santiago
- Croatia (5):
  - General Hospital Karlovac, Karlovac
  - Thalassotherapia, Opatija
  - KBC Split, Split
  - Clinical Hospital "Sveti Duh", Zagreb
  - University Hospital Sisters of Mercy, Zagreb
- France (10):
  - CHU Avicenne, Bobigny
  - Hopital Pellegrin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Bicêtre, Université Paris-Sud 11, INSERM U802, Le Kremlin-Bicêtre
  - C.H.U. Hôpital Roger Salengro, Lille
  - Hôpital Lapeyronie, Montpellier
  - Hôpital Xavier Bichat, Paris
  - Hopital La Pitie Salpetriere, Paris
  - Hopital Lariboisière, Paris
  - CHU Strasbourg-Hautepierre, Strasbourg
- Romania (4):
  - "Dr. Constantin Opris" Emergency County Hospital Baia Mare, Baia Mare
  - "Dr. I Cantacuzino" Clinical Hospital, Bucharest
  - Ianuli Med Consult SRL, Bucharest
  - Rehabilitation Clinical Hospital Iasi, Iași

REFERENCES:
- [Derived] Durez P, Vandepapeliere P, Miranda P, Toncheva A, Berman A, Kehler T, Mociran E, Fautrel B, Mariette X, Dhellin O, Fanget B, Ouary S, Grouard-Vogel G, Boissier MC. Therapeutic vaccination with TNF-Kinoid in TNF antagonist-resistant rheumatoid arthritis: a phase II randomized, controlled clinical trial. PLoS One. 2014 Dec 17;9(12):e113465. doi: 10.1371/journal.pone.0113465. eCollection 2014. PMID 25517733